CLINICAL TRIAL: NCT03063593
Title: UK Multi-Centre, Observational, Post-Market Clinical Follow-up of the INFINITY® Total Ankle System
Brief Title: UK Infinity, Post-Market Clinical Follow-up Study
Status: Active, not recruiting | Type: Observational
Sponsor: Stryker Trauma and Extremities (Industry)
Responsible Party: Sponsor
Other Study IDs: UK15-TAR-001
Record Dates: First submitted 2017-02-15; First posted 2017-02-24 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Arthritis, Rheumatoid; Post-traumatic Osteoarthritis; Degenerative Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study Title UK Post-Market Clinical Follow-Up Of The INFINITY® Total Ankle System Study Design Prospective, multi-site, multi-year post-market clinical follow-up study Study Group Primary/Unilateral and/or bilateral Total Ankle Arthroplasty subjects implanted with INFINITY® Total Ankle System Number of Subjects 500 with 10 sites

DETAILED DESCRIPTION:
Study Title UK Post-Market Clinical Follow-Up Of The INFINITY® Total Ankle System Study Design Prospective, multi-site, multi-year post-market clinical follow-up study Study Group Primary/Unilateral and/or bilateral Total Ankle Arthroplasty subjects implanted with INFINITY® Total Ankle System N Subjects 500 with 10 sites Follow-Up Schedule Subject enrollment will consist of a Pre-operative, Operative, 6 months, 1 yr., 2 yr., 5yr., 7 yr., 10 yr., and an unscheduled visit as needed.

Primary Objective Evaluate the long-term survivorship of the INFINITY® implant over 10 years

Secondary Objective(s) Secondary objectives assessed will be to:

* Identify and assess the implant for component loosening and/or subsidence, any osteolysis and/or cyst formation through radiographic evaluation early and throughout the lifetime of the implant.
* Compare the improvements in self-reported pain and social interaction for quality of life measures from pre-op through 10 years post operatively; assessed by EuroQol (EQ5D5L).
* Compare pain and functional improvement in the Ankle Osteoarthritis Score (AOS), which is a visual analogue scale specifically designed as a modification of the Foot Function Index.
* Compare the improvement in self-reported pain-free function scores from pre-op through 10 years post-operatively, assessed by the Manchester Oxford Foot Questionnaire (MOXFQ) walking/standing scores.
* Identify and report the safety of the implant in terms of complications and adverse events.

Inclusion Criteria Subjects to be included in the study must meet all of the following criteria:

* Be 21 years of age at the time of surgery;
* Diagnosed with unilateral and/or bilateral ankle joint disease;
* Diagnosed with ankle joint damage from rheumatoid arthritis, post-traumatic, or degenerative arthritis; Willing and able to consent to participate (written, informed consent / witnessed verbal consent) Willing and able to attend the requested follow-up visits;
* Subjects determined by the Investigator to be an appropriate candidate for the INFINITY® Total Ankle System

Exclusion Criteria Subjects will be excluded from the study if they meet any of the following criteria:

* Subjects with an ankle condition, as determined by the investigator, to be an inappropriate candidate for a total ankle replacement;
* Subjects requiring revision total ankle replacement of the ankle being considered for study

ELIGIBILITY:
Inclusion Criteria:

Subjects to be included in the study must meet all of the following criteria:

* Be 21 years of age at the time of surgery;
* Diagnosed with unilateral and/or bilateral ankle joint disease;
* Diagnosed with ankle joint damage from rheumatoid arthritis, post-traumatic, or degenerative arthritis; Willing and able to consent to participate (written, informed consent / witnessed verbal consent) Willing and able to attend the requested follow-up visits;
* Subjects determined by the Investigator to be an appropriate candidate for the INFINITY® Total Ankle System

Exclusion Criteria:

Subjects will be excluded from the study if they meet any of the following criteria:

* Subjects with an ankle condition, as determined by the investigator, to be an inappropriate candidate for a total ankle replacement;
* Subjects requiring revision total ankle replacement of the ankle being considered for study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Primary/Unilateral and/or bilateral Total Ankle Arthroplasty subjects implanted with INFINITY® Total Ankle System
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-04-29 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure survivorship at 10 years | 10 Years
  The primary outcome measure of this post-market clinical observational study is to collect data relating to the INFINITY® Total Ankle System performance/survivorship at up to 10 years.

SECONDARY OUTCOMES:
EQ5D-EuroQol-questionnaire | From pre-op through 10 years
  Compare the improvement in self-reported pain and social interaction for quality of life measures
Ankle Osteoarthritis Score (AOS)-questionnaire | From Pre-op through 10 years
  Self-reported to compare pain and functional improvement, which is a visual analogue scale specifically designed as a modification of the Foot function Index
Manchester Oxford Foot Questionnaire (MOXFQ)-questionnaire | From Pre-op through 10 years
  Compare the improvement in self-reported pain-free function scores (walking/standing scores)
Radiographic evaluation-physician reported questionnaire | From Pre-op through 10 years
  identify and assess the implant for component loosening and/or subsidence, any osteolysis and/or cyst formation

CONTACTS AND LOCATIONS:
Overall Officials: David Townshend, MD, Study Chair — Northumbria Trust; Rebecca Gibson, Study Director — Stryker Trauma & Extremeties
Locations (12):
- United Kingdom (12):
  - Torbay Hospital, Torquay, Devon
  - Royal Bournemouth Hosptial, Bournemouth, Dorset
  - University Hairmyres Hospital, Bothwell, Scotland
  - RJAH Orthopaedic Hospital, Oswestry, Shropshire
  - Sheffield Teaching Hospital, Sheffield, South Yorksire
  - North Bristol NHS Trust Southmead Hospital, Bristol
  - Royal Infirmary of Edinburgh, Edinburgh
  - Royal Devon and Exeter NHS Foundation Trust, Exeter
  - Royal National Orthopaedic Hospital, Middlesex
  - North Tyneside General Hospital, Newcastle upon Tyne
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Wrightington Hospital, Wigan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2017-10-06): https://cdn.clinicaltrials.gov/large-docs/93/NCT03063593/Prot_000.pdf